Focus of attention in individuals post-stroke

Focus of attention effects on motor performance and learning in individuals post stroke during seated lateral weight shifting: A feasibility study

December 21, 2020

Ashley Watamura Hyatt, PT, DPT, NCS Assistant Professor Department of Physical Therapy Western Carolina University 3971 Little Savannah Road Cullowhee, NC 28723 awhyatt@email.wcu.edu

Ann Medley, PT, PhD
Professor, Director
School of Physical Therapy
Texas Woman's University
5500 Southwestern Medical Ave.
Dallas, TX 75235-7299
smedley@twu.edu

## Corresponding author:

Ashley Watamura Hyatt, PT, DPT, NCS, 3971 Little Savannah Road, Cullowhee, NC 28723, 717-682-9710, <a href="mailto:awhyatt@email.wcu.edu">awhyatt@email.wcu.edu</a>

The authors have no conflict of interest to declare.

Keywords: Stroke, focus of attention, motor learning, seated weight shifting

IRB approval:

Western Carolina University, reference number 949671-4 Mission Health, reference number 1124795-3

# Western Carolina University College of Health and Human Sciences Department of Physical Therapy

### **Informed Consent for Participation in Research Study**

The Impact of Instructional Strategies on Seated Trunk Control in Healthy Adults and Adults Post Stroke: A Motor Learning Study

This study will help us understand which instructions work best when teaching adults how to enhance their seated balance. Your participation in this study may ultimately enhance your balance during everyday tasks that often occur while sitting.

## Description of the research and your participation

## **Time requirements**

You will be asked to participate in one one-hour session including time for completion of pre and post training tasks and instruments. We would like for you to return one week later for a follow up session in order to run a few of the tasks again. This final session should last about 30 minutes.

### Risks and discomforts

No known risks are associated with this research. Vitals will be monitored and a licensed physical therapist will be present during all sessions. The task may be strenuous at times depending on your physical abilities, but rest breaks will be provided as necessary.

#### **Potential benefits**

Your sitting balance may improve with this training both in a still position and with movement.

### **Protection of confidentiality**

We will do everything we can to protect your privacy. Only the research team will have access to your information relevant to the data being collected. Your identity will not be revealed in any publication that might result from this study. With your permission, you may be video recorded during your session to accurately collect data to evaluate the effectiveness of the training you received. Your name, voice, and personal information will not be recorded on the video and confidentiality will be strictly maintained.

# Voluntary participation

Your participation is completely voluntary. You may choose not to participate and withdraw from the study at any time. Your information, including your responses to the survey and your performance will be kept anonymous.

#### **Contact Information**

If you have questions about this study, contact Dr. Ashley Hyatt at the Department of Physical Therapy, Western Carolina University, Cullowhee, NC 28723 (828-227-2296). If you have any questions or concerns about your treatment as a participant in this study, you can reach the Chair of the Western Carolina University Institutional Review Board through WCU's Office of Research Administration at 828-227-7212.

#### Consent

| I am at least 18 years of age and have read this consent form and have been given | the |
|---|---|
| opportunity to ask questions. I give my consent to participate in this study. | |

| Participant's signature: | Date: |
|-------------------------------------|-------|
| Assistant investigator's signature: | Date: |

At least one of the following researchers listed above will read this consent form to you and serve as a witness. A copy of this consent form should be given to you.

# Permission Form for Photography/Video in a Research Study Western Carolina University

With your permission, you will be photographed/videotaped during this study. Your name, voice, or personal information will not be recorded on the image and confidentiality will be strictly maintained.

Photographs or video taken during this study for the purpose of collecting data and presenting findings for educational purposes will be maintained electronically on a password protected computer for a period of 10 years. After this time period, electronic files will be destroyed.

If you desire to participate and be photographed/videotaped, please sign the following statement that indicates your permission to use the photograph/video. You will be provided opportunity after the recording to refuse your participation if the image is not to your liking.

| | ed/videotaped for this project and for th<br>uals regarding the outcomes of this study | |
|---|---|---|
| Signature of Volunteer | Date | |
| 0 ' | ained to the participant the purpose, the sk of this photograph/video; and the alte | ernatives to |
| Signature of Researcher | Date | |